CLINICAL TRIAL: NCT06454877
Title: Effect of Normothermia Care Bundle on Inadvertent Perioperative Hypothermia, Surgical Site Infection and Bleeding in Knee Replacement Surgery
Brief Title: Effect of Normothermia Care Bundle in Knee Replacement Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Saglik Bilimleri University (Other)
Responsible Party: Principal Investigator, Gulsen Ozturk Genc, PhD Student, Istanbul Saglik Bilimleri University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IstanbulSBU-OZTURKGENC-001
Record Dates: First submitted 2024-06-04; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Knee Prosthesis
Keywords: Hypotermia; surgical site infection; active heating; pasive heating; nursing care bundle
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- active heating (Experimental): It is the group to be actively heated with the heating method using hot air blowing device.
  Interventions: Device: active heating
- pasive heating (Experimental): Passive heating using reflective blankets is the group to be made.
  Interventions: Behavioral: pasive heating
- control group (No Intervention): The group will receive routine hospital care without any intervention.

INTERVENTIONS:
Device: active heating — Preheating will be performed for 15 minutes 30 minutes before surgery with a hot air blowing device in accordance with the normothermia care package so that the body temperature is 36-37 C°.
  Active heating during surgery will be done with a heating bed placed on the operating table.
  Patients taken to the postoperative care unit will continue to be heated with a hot air blower and the device will be turned off when the body temperature reaches 37 C°.
  Arms: active heating
Behavioral: pasive heating — In accordance with the normothermia care package, the reflective blanket will be covered to cover the whole body 30 minutes before surgery.
  During the operation, the body will be covered with a reflective blanket in accordance with the surgical intervention.
  Patients taken to the postoperative care unit will continue to be warmed with reflective blankets.
  Arms: pasive heating

SUMMARY:
Osteoarthritis is a disease characterized by disruption of the integrity of articular cartilage as a result of erosion of articular cartilage. Knee osteoarthritis causes muscle weakness, crepitation and deformities in the knee joint, limiting the individual's movement and causing loss of function. The most prominent feature is pain. Therefore, knee replacement surgery is performed in advanced cases where pharmacologic treatment is not effective. Many complications can be seen during the operation process and some of them may occur due to hypothermia. Studies have reported that warming during the operation prevents hypothermia and reduces complications. In this study, it was aimed to examine the effect of active and passive heating applied before, during and after surgery on hypothermia, surgical site infections and bleeding. The population of the study will consist of patients who underwent knee replacement surgery in the Orthopedics and Traumatology Clinic of Üsküdar State Hospital between April 2024 and April 2025. Data will be collected using the patient identification form, normothermia care package observation form, preoperative follow-up form, postoperative follow-up form and postoperative long-term follow-up form. A randomization list generated from a computer-based random numbers table will be used to determine which group of patients will be included in the study. Patients will be followed up in 3 periods: preoperative, intraoperative and postoperative periods. The postoperative period will be evaluated in five stages as day 1, day 2, day 3, day 10 and day 30. The purpose of the study and the intervention to be applied will be explained to all groups to be included in the study by the researcher and written and verbal consent will be obtained from the volunteers. The groups included in the study will be subjected to the heating protocol according to the normothermia care package. Group A will receive active heating with the heating method using a hot air blowing device. Group B will receive passive heating using a reflective blanket. Group C was planned as a control group to be heated by applying the routine heating procedure of the hospital without any intervention. Body temperature and vital signs will be checked preoperatively and warming will be performed 30 minutes before surgery, and warming will be started 15 minutes before anesthesia induction during surgery and body temperature and vital signs will be checked. After the operation and in the ward, warming will be performed until the body temperature reaches 37 C°. The data obtained will be analyzed using SPSS (Statistical Package for Social Sciences) for Windows 22.0 program.

ELIGIBILITY:
Inclusion Criteria:

18 years or older Planned elective knee arthroplasty surgery Patients planned for neuraxial block anesthesia ASA (American Society of Anesthesiologists) class I-III

Exclusion Criteria:

Alcohol and drug addiction, Patients who cannot be contacted Preoperative body temperature <36 C° or ≥37.5 C°

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
vital signs observation form | Before surgery, during surgery, first 24 hours after surgery and first 3 days after surgery
  in this form body temperature value will be evaluated
vital signs observation form | Before surgery, during surgery, first 24 hours after surgery and first 3 days after surgery
  In this form, diastolic and systolic blood pressure will be evaluated
vital signs observation form | Before surgery, during surgery, first 24 hours after surgery and first 3 days after surgery
  in this form thermal comfort score will be evaluated. Thermal comfort scale evaluation will be evaluated with a visual analog scale. It is a scale with 10 points at one end of the scale and 100 points at the other end. The patient will be asked to mark his/her comfort level.
vital signs observation form | Before surgery, during surgery, first 24 hours after surgery and first 3 days after surgery
  in this form level of tremor will be evaluated.The tremor level evaluation form is evaluated between 0-3. 0 points: no tremor, 1 Mild: tremor localized only in the neck and/or thorax, 2 Moderate: tremor in the neck, thorax and upper extremities, 3 Severe: It is evaluated as tremors in the trunk, upper and lower extremities.
vital signs observation form | Before surgery, during surgery, first 24 hours after surgery and first 3 days after surgery
  in this form heart rate will be evaluated

SECONDARY OUTCOMES:
bleeding follow-up form | first 3 days after surgery
  Hb (hemoglobin) will be evaluated in terms of bleeding.
bleeding follow-up form | first 3 days after surgery
  Hct (Hemotocrit)will be evaluated in terms of bleeding.
bleeding follow-up form | first 3 days after surgery
  PT(Protrombin time) will be evaluated in terms of bleeding.
drain follow-up form | first 3 days after surgery
  the amount of drainage will be evaluated for bleeding
observation form assessing surgical site infection | To be evaluated on the 3rd day, 10th day and 30th day after surgery
  WBC (White Blood Count) will be evaluated for surgical site infection
observation form assessing surgical site infection | To be evaluated on the 3rd day, 10th day and 30th day after surgery
  CRP (C Reaktif Protein)will be evaluated for surgical site infection
observation form assessing surgical site infection | To be evaluated on the 3rd day, 10th day and 30th day after surgery
  will be evaluated for surgical site infection